CLINICAL TRIAL: NCT03904784
Title: School Withdrawal in Adolescents: Impact of the Ambulatory Child Psychiatry Therapeutic Device. Prospective Study
Brief Title: School Withdrawal in Adolescents
Acronym: DESCOL
Status: Terminated | Type: Observational
Why Stopped: During the pandemic covid-19 the school is not in the classroom
  The study cannot continue
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Other Study IDs: DESCOL
Record Dates: First submitted 2019-04-04; First posted 2019-04-05 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-06

CONDITIONS: Depression; Anxiety Disorders; Obsessive-Compulsive Disorder; Behavior Disorders; Emotional Disorder; Somatoform Disorders; Neurotic Disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Obsessive-Compulsive Disorder; Mental Disorders; Somatoform Disorders; Neurotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- School withdrawal teenagers: The study is based on questionnaries, interview with teenagers and/or their familly
  Interventions: Behavioral: school withdrawal teenagers

INTERVENTIONS:
Behavioral: school withdrawal teenagers — The teenagers will have 4 interview with medical team alone or with his familly in order to have questionnaries, schools reports, psychological evaluation.

SUMMARY:
The aim of the study is to evaluate the impact of the outpatient ambulatory child psychiatric care system on the functioning of anxio-depressive adolescents in school retreat by describing the modalities of individual psychic functioning.

DETAILED DESCRIPTION:
This research project concerns adolescent patients aged 12 to 17, a period of life towards psychic individualization and autonomy. It is part of an outpatient child psychiatry sector that is concerned with the multidisciplinary and institutional dimension of the care provided. These are part of a long-term patient care dynamic. It is a therapeutic accompaniment of the young person and his entourage, especially parents.

The care is integrative and multidisciplinary (psychiatrist, psychologist, educator, psychomotor, nurse). The care project is done after team discussion, several points are taken into account (clinical evaluation, demand analysis, transfer, study of different psychic movements, family dynamics). The eyes are crossed and the various references (psychodynamic, psychoanalytic, systemic). The family consultations that are always present can be associated with the individual care of the young person, and always link with the analysis of the different institutional movements. This takes place especially at the time of the weekly clinical summaries where the clinical situations of concern are evoked to allow a cross reading and multidisciplinary.

The reflection, the exchange between the various stakeholders allow to weave an institutional mesh containing. Thanks to this system, young people and their families can experience a continuous and solid relationship.

The sector is also part of a very valuable network work with the various partners involved in the daily life of the young person and their family (school institution, social services ...).

This research is intended to be as close as possible to the care we provide and is integrated into a global work whose main interest is that of the patient.

ELIGIBILITY:
Inclusion Criteria:

* New patients in the sector with a problem of school withdrawal previously educated in ordinary medium without MDPH file (Departmental House of Disabled People).
* Young people out of school: school attendance less than 50% of school time for one month (absent at least half of school time)
* Clinical diagnosis according to the International Classification of Diseases 10 (ICD 10): F32 (depressive episodes), F33 (recurrent depressive disorder), F40 (phobic anxiety disorders), F41 (other anxiety disorders), F42 (obsessive-compulsive disorders), F43 (reaction to severe stressor, and adjustment disorders), F45 (somatoform disorder), F48 (other neurotic disorders), F90 to F98 Behavioral and emotional disorders usually occurring during childhood and adolescence
* Accepting to participate in the clinical research device

Exclusion Criteria:

* Other psychiatric diagnoses (schizophrenia, BDA (acute delirious puff), TED (Invasive Disorder of Development)).
* Intellectual deficit proved
* Education in SEGPA (Section of General and Adapted Professional Education) and ULIS (Localized Unit for School Inclusion)
* Somatic illness preventing attendance at a school
* Refusal to participate in the study

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: teenagers between 12 and 17 years who are anxio-depressive and school retreat
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
psychological assessment | 18 months
  interview of the teenager with a psychologist

SECONDARY OUTCOMES:
school report | 18 months
  change in school level
familly questionnary | 18 months
  interview of the family with a psychologist

CONTACTS AND LOCATIONS:
Locations (1):
- 1er secteur de psychopathologie de l'enfant et de l'adolescent du Val de Marne, Champigny-sur-Marne, France

IPD SHARING:
Plan to Share IPD: No